CLINICAL TRIAL: NCT05524220
Title: Effect of Nasal Positive Airway Pressure Versus Standard Care on Oxygenation and Ventilation During Propofol-based Sedation for Colonoscopy in Patients With High Risk of Airway Obstruction: a Prospective Randomized Controlled Trial.
Brief Title: Effect of Nasal Positive Airway Pressure Versus Standard Care on Oxygenation and Ventilation During Propofol-based Sedation for Colonoscopy in Patients With High Risk of Airway Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Vyaire Medical (Industry)
Responsible Party: Principal Investigator, Erikka L Washington, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0351
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea, Obesity
Keywords: Obstructive Sleep Apnea; total IV anesthesia; obesity; colonoscopy; Nasal cpap
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: Standard care with a facemask. (Active Comparator)
  Interventions: Device: Standard care with a facemask.
- Group B: SuperNO2VA™EtCO2 (Experimental)
  Interventions: Device: SuperNO2VA™EtCO2 (Nasal Oxygenating Ventilating Apparatus)

INTERVENTIONS:
Device: Standard care with a facemask. — The anesthesia provider will supply oxygen via the closed facemask at 10 liters per minute (LPM)
  Arms: Group A: Standard care with a facemask.
Device: SuperNO2VA™EtCO2 (Nasal Oxygenating Ventilating Apparatus) — The anesthesia provider will attach the SuperNO2VA™ EtCO2 circuit port to the hyperinflation bag with the oxygen flow rate to 10 L/min. The oxygenation, continuous positive airway pressure, and ventilation of the subject will be done via SuperNO2VA™EtCO2 (Nasal Oxygenating Ventilating Apparatus)
  Arms: Group B: SuperNO2VA™EtCO2

SUMMARY:
The purpose of this study is to to compare oxygenation and ventilation on spontaneously ventilating obese patients or those with diagnosed or undiagnosed Obstructive sleep apnea (OSA) undergoing day colonoscopy under Propofol based sedation, between the SuperNO2VA Et™ nasal positive airway pressure (PAP) device and routine care with face mask for oxygen (O2).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy
* American Society of Anesthesiology (ASA) Physical Status I-III
* BMI ≥30 kg/m2 or suspected Obstructive Sleep Apnea

Exclusion Criteria:

* Inpatient status
* Active Congestive Heart Failure Exacerbation
* Untreated ischemic heart disease
* Acute exacerbation of respiratory disorders, including Chronic obstructive pulmonary disease (COPD) and asthma
* Emergent procedures
* Pregnancy
* Previous enrollment in this study
* Inability to provide informed consent
* Additional medical testing planned for the same day
* History of allergic reaction to Propofol
* Tracheostomy
* Supra-glottic or sub-glottic tumor
* Gastrointestinal tract obstruction or delayed transit (including delayed gastric emptying, gastric bezoar, achalasia, toxic megacolon).
* Prisoners
* Unable to fit SuperNoVa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erikka Washington, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Started | 71 | 68
Completed | 71 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask. | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [51 to 64] | 54.5 [48.5 to 62] | 56 [50 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 90
  Male | 25 | 24 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 45 | 93
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 52 | 107
  Black or African-American | 15 | 15 | 30
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 71 | 68 | 139
American Society of Anesthesiology (ASA) Classification [Count of Participants; unit: Participants] — ASA Physical Status Classification System - The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I :A normal healthy patient ASA II :A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes Population: Data were not collected from 1 participant in the Group B: SuperNO2VA™EtCO2 arm.
  Participants
    number analyzed (Participants) | 70 | 68 | 138
    ASA I: A normal healthy patient | 0 | 0 | 0
    ASA II: A patient with mild systemic disease | 19 | 21 | 40
    ASA III: A patient with severe systemic disease | 51 | 47 | 98
    ASA IV: A patient with severe systemic disease that is a constant threat to life | 0 | 0 | 0
    ASA V: A moribund patient who is not expected to survive without the operation | 0 | 0 | 0
    ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes | 0 | 0 | 0
Body Mass Index [Median (Inter-Quartile Range); unit: kilograms per square meter] | 36.6 [32.5 to 40.9] | 35.2 [33.5 to 39.7] | 35.9 [32.7 to 40.3]
Body Mass Index [Count of Participants; unit: Participants]
  < 30 | 1 | 2 | 3
  30 ≤ BMI < 40 (obesity) | 50 | 49 | 99
  ≥ 40 (Class 3 obesity) | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Time Taken From Initiation of Induction to the First Airway Intervention
Time Frame: From Initiation of Induction to the First Airway Intervention (about 16 minutes)
Population: 16 participants in the Group B: SuperNO2VA™EtCO2 needed airway intervention. 29 participants in the Group A: Standard care with a facemask needed airway intervention. Only the participants who needed airway intervention were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 16 | 29
minutes | 5 [3 to 11] | 10 [4.5 to 15.5]

2. Secondary Outcome: Amount of Propofol Administered During Induction
Time Frame: Within 5 minutes of the start of anesthesia
Measure: Mean (Inter-Quartile Range); unit: milligrams
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
milligrams | 70 [50 to 100] | 75 [50 to 100]

3. Secondary Outcome: Total Amount of Propofol Administered During the Procedure
Time Frame: during the procedure (about 45 minutes)
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
milligrams | 360 [220 to 450] | 253 [200 to 455]

4. Secondary Outcome: Change in Alertness of Subject as Assessed by the Modified Observer's Assessment of Alertness/Sedation Scale (MOAAS)
Description: This is scored from 0(no response)-5(response to your name spoken in a normal tone), a higher number indicating more alertness
Time Frame: prior to endoscopic intubation,during the procedure
Population: Data were not collected for this outcome measure because the assessment was not done by the observers. As a result, 0 observers completed the assessment, and therefore, no participants were analyzed in either study arm.
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time Taken From Induction to Endoscopic Insertion
Time Frame: within 10 minutes of start of sedation
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
minutes | 2 [2 to 4] | 3 [2 to 9]

6. Secondary Outcome: Incidence of Procedural Interruptions as Assessed by the Number of Times the Endoscope is Removed From the Patient
Time Frame: From Initiation of Induction to removal of endoscope at the end of the procedure (about 45 minutes)
Measure: Number; unit: number of times endoscope is removed
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
number of times endoscope is removed | 0 | 0

7. Secondary Outcome: Duration of Procedural Interruptions as Assessed by the Length of Time the Endoscope is Removed From the Patient
Time Frame: From Initiation of Induction to removal of endoscope at the end of the procedure (about 45 minutes)
Population: Zero participants had a procedural interruption.
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Received Airway Maneuvers
Time Frame: From Initiation of Induction to removal of endoscope at the end of the procedure (about 45 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
Participants | 16 | 29

9. Secondary Outcome: Time Taken for Airway Maneuvers
Time Frame: From Initiation of Induction to removal of endoscope at the end of the procedure (about 45 minutes)
Population: 16 participants who received airway maneuvers in the Group B: SuperNO2VA™EtCO2 arm were analyzed for the outcome measure. 29 participants who received airway maneuvers in the Group A: Standard care with a facemask arm were analyzed for the outcome measure.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 16 | 29
seconds | 172.5 [39.5 to 1247] | 131 [33 to 621]

10. Secondary Outcome: Reason for Airway Maneuvers
Time Frame: From Initiation of Induction to removal of endoscope at the end of the procedure (about 45 minutes)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 16 | 29
Participants
  Apnea | 2 | 9
  Desaturations <90% SpO2 | 12 | 10
  Apnea and Desaturations <90% SpO2 | 2 | 9
  Other | 0 | 1

11. Secondary Outcome: Time Taken for the Entire Procedure
Time Frame: from start of procedure to end of procedure (about 45 minutes)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
minutes | 33 [29 to 44] | 33.5 [26 to 40.5]

12. Secondary Outcome: Recovery Time as Assessed by the Time When Subject Was Ready for Discharge
Time Frame: at time of discharge( about one hour from end of procedure)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
minutes | 48 [36 to 57] | 46.5 [33 to 56.5]

13. Secondary Outcome: Recovery Time as Assessed by the Actual Time When Subject Was Discharged
Time Frame: at time of discharge( about one and a half hour from end of procedure)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
minutes | 81 [70 to 96] | 77 [66 to 92.5]

14. Secondary Outcome: Patient Satisfaction as Assessed by the Visual Analog Scale (VAS)
Description: This will be scored from 0-10, a higher score indicating more satisfaction
Time Frame: at time of discharge(about one hour from end of procedure)
Population: Data were not collected from 3 participants in the Group B: SuperNO2VA™EtCO2 arm because the participants did not complete the survey. Data were not collected from 1 participant in the Group A: Standard care with a facemask arm because the participant did not complete the survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 68 | 67
score on a scale | 10 [10 to 10] | 10 [10 to 10]

15. Secondary Outcome: Number of Participants That Tolerated the SuperNO2VA™EtCO2
Time Frame: from start of procedure to end of procedure (about 45 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Group B: SuperNO2VA™EtCO2
Number analyzed (Participants) | 71
Participants | 69

16. Secondary Outcome: Anesthesiologist Satisfaction Score as Assessed by the Visual Analog Scale (VAS)
Description: This will be scored from 0-10, a higher score indicating more satisfaction
Time Frame: end of procedure (about 45 minutes from start)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
score on a scale | 8.5 [7 to 10] | 8 [7 to 10]

17. Secondary Outcome: Number of Participants That Had Incidences of Cardiac Complications
Time Frame: during the procedure (about 45 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
Number analyzed (Participants) | 71 | 68
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to discharge (up to 24 hours)
Arm/Group | Group B: SuperNO2VA™EtCO2 | Group A: Standard Care With a Facemask.
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group B: SuperNO2VA™EtCO2 (N=71) | Group A: Standard Care With a Facemask. (N=68)
needed supplemental oxygen after procedure (Injury, poisoning and procedural complications) | 1 | 0
concern for bleeding after polyp removal (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT05524220/Prot_SAP_000.pdf